CLINICAL TRIAL: NCT01072370
Title: A Placebo-Controlled, Observer-Blinded, Crossover Study to Evaluate the Safety and Effectiveness of a Single, Autologous, Cord Blood Stem Cell Infusion for the Treatment of Cerebral Palsy in Children
Brief Title: Safety and Effectiveness of Cord Blood Stem Cell Infusion for the Treatment of Cerebral Palsy in Children
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, James E. Carroll, Professor and Chief, Child Neurology, Augusta University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACBSC09
Record Dates: First submitted 2010-02-16; First posted 2010-02-22 (Estimated); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Cerebral Palsy
Keywords: Umbilical Cord Blood; Stem Cells; Autologous Blood Transfusion; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group 1 (Active Comparator)
  Interventions: Biological: Cord Blood Infusion
- Treatment Group 2 (Sham Comparator)
  Interventions: Biological: Intravenous Sham

INTERVENTIONS:
Biological: Cord Blood Infusion — red-cell depleted, mononuclear cell enriched cord blood unit prepared for infusion
  Other Names: Stem cell infusion
  Arms: Treatment Group 1
Biological: Intravenous Sham — intravenous infusion of 5% dextrose, ¼ normal saline solution
  Other Names: Placebo
  Arms: Treatment Group 2

SUMMARY:
The purpose of this study is to test the safety and effectiveness of a cord blood infusion in children who have motor disability due to cerebral palsy (CP). The subjects will be children whose parents have saved their infant's cord blood, who have non-progressive motor disability, and whose parents intend to have a cord blood infusion.

DETAILED DESCRIPTION:
The purpose of this study is to conduct an observer-blinded crossover investigation of the safety and efficacy of autologous cord blood infusion in children who demonstrate non-progressive motor disability due to brain dysfunction (commonly called cerebral palsy) and who do not have an apparent disorder of brain development or obstructive hydrocephalus. The degree of delay in motor development will be such that the children are unable to sit independently by 12 months of age or unable to walk independently by 18 months of age. However, because the diagnosis is one of exclusion, we will enroll patients only after they have reached two years of age. By this age, it is likely other conditions would be excluded. As the Gross Motor Function Classification System (GMFCS) was developed for children up to 12 years of age, the maximum age of recruitment will be 12 years. Any level of cerebral palsy severity will be allowed. The subjects will be children whose parents have saved their infants cord blood, who have clinical evidence of a non-progressive motor disability, and whose parents intend to have a cord blood infusion.

ELIGIBILITY:
Inclusion Criteria:

* Must be more than 1 year of age and less than 12 years of age at the time of screening for inclusion in the study.
* Clinical evidence of a non-progressive motor disability due to brain dysfunction. The subjects will not have the ability to sit independently by one year of age or the ability to walk by 18 months of age.
* Have stored umbilical cord blood with Cord Blood Registry (CBR) that meets all selection and testing criteria.
* Willing to comply with all study procedures.
* The nucleated cells available in the cord blood sample stored at CBR must exceed 1 X 107 cells per kg body weight. (Note: Because cord blood collection has been in process for about 16 years but widely for far less than that period, the age of most subjects likely will be considerably less than 12 years of age. Due to the amount due of cord blood available for most subjects, the body weight of subjects usually will not exceed 25 kg).
* The patients must be seizure-free or seizures adequately controlled. If there is a suspicion of seizures and EEG should be done prior to inclusion.

Exclusion Criteria:

* Have complicating medical issues that would interfere with blood drawing, such as venous access so limited that success is unlikely
* Presence of obstructive hydrocephalus.
* Presence of progressive neurological disease.
* Presence of significant defect of brain development, such as schizencephaly or agenesis of corpus callosum
* Presence of known chromosomal anomaly
* Presence of major congenital anomaly
* Severe intrauterine growth restriction (birth weight less than 1800 grams)
* Cord blood viability <60%
* Positive infectious disease markers from mother's blood or cord blood at the time of collection.
* Evidence of illness on planned infusion date (such as but not limited to fever >38.5, vomiting, diarrhea, wheezing, or crackles)
* Pregnancy
* Use of immunosuppressive drugs
* Evidence of known genetic disorder
* Impaired hepatic or renal function

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Confirm the safety of autologous cord blood infusion in children with cerebral palsy by repeated follow-up over one year with clinical and laboratory evaluations. | 1 year

SECONDARY OUTCOMES:
Confirm the efficacy of autologous cord blood infusion in children with cerebral palsy using patient questionnaire and standardized Gross Motor Function Measure evaluation. | 3-4 months

CONTACTS AND LOCATIONS:
Overall Officials: James E Carroll, M.D., Study Chair — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

REFERENCES:
- See also: Augusta University — http://www.augusta.edu